CLINICAL TRIAL: NCT04120935
Title: A Master Protocol Empowering Precision Research in Colorectal Cancer
Brief Title: ALFAOMEGA Master Observational Trial
Acronym: ALFAOMEGA
Status: Recruiting | Type: Observational
Sponsor: IFOM ETS - The AIRC Institute of Molecular Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IFOM-CPO003/2018/PO002
Record Dates: First submitted 2019-09-18; First posted 2019-10-09 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * FFPE Tissue
  * Fresh Tissue (tumor and normal)
  * Plasma
  * PBMC
  * Whole Blood
  * Stools
  * Buccal Swabs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort of CRC patients: Stage-mixed cohort of at least 3000 patients through their course of treatments, until death or a minimum of 5 years.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Prospective Observation of standard clinical practice.

SUMMARY:
AlfaOmega has been designed to streamline the study of the co-evolutionary landscape between tumor and host cells in a cohort of CRC patients, with the aim of understanding how their outcomes can be significantly improved (e.g. reduction of their chance of recurrence and survival improval). This clinical resource for integrative clinical data and sample collection will allow the molecular story-telling of CRC metastatic spread along time and space and the selection of appropriate patients for experimentally-driven trials.

DETAILED DESCRIPTION:
AlfaOmega is an observational study that will follow a stage-mixed cohort of at least 500 patients through their course of treatments, until death or a minimum of 5 years. Patients will be longitudinally sampled and matched clinical data (including imaging) will be collected. Via a multi-tiered informed consensus process, AlphaOmega will also allow to develop companion diagnostics for molecular enrichment strategies in AIRC-driven proof-of-concept trials. To achieve the required level of 'experimental precision', patients will enter AlphaOmega at two different 'therapeutic checkpoints': i) prior to a surgical event or ii) prior to a systemic treatment. In the latter case patients with no previous lines of therapy for metastatic disease will be privileged.

To optimize the enrollment of patients, the longitudinal collection of data/samples and their logistic management, AlphaOmega has been designed as a flexible infrastructure organized in TIERS for the stepwise comprehension of the biological processes that drive tumor evolution, and precisely:

* TIER1, Monitoring: the ability to follow CRC evolution under standard of care treatments and to define new evolution-linked biomarkers. This will be achieved through the collection of clinical data, imaging data, FFPE tissue and frozen plasma/PBMC.
* TIER2, Modelling: the ability to develop pertinent experimental models to study evolutionary mechanisms and define evolution-targeting therapeutic strategies. This will be achieved through the collection of Fresh Tissue, Whole Blood, Stools, Buccal Swabs and other fluids.
* TIER3, Linking: the ability to access data and samples of patients enrolled in proof-of-concept trials to prove the efficacy and study/understand resistance mechanisms of evolution-targeting therapies. This will be achieved by introducing the connection in the trial protocol.

ELIGIBILITY:
Inclusion Criteria:

1. TIER1 written Informed consent.
2. Patients ≥18 years of age.
3. Previous diagnosis of colorectal cancer, or a strong suspicion of CRC based on clinical and radiological findings.
4. In patients with previous diagnosis of CRC availability of diagnostic Formalin-Fixed, Paraffin Embedded (FFPE) blocks (surgical resection and/or tumor biopsies), or at least 10 slides (preferably 20). FFPE tissue blocks are always preferred to slides.
5. ECOG Performance status < 2.

Exclusion Criteria:

1. Any other current malignancy or malignancy diagnosed or relapsed within the past 5 years (other than non-melanomatous skin cancer, stage 0 melanoma in situ, and in situ cervical cancer)
2. Patient unable to comply with the study protocol owing to psychological, social or geographical reasons.
3. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or syphilis infection.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients longitudinally monitored | 6 months
  1. - Number of recruited CRC cases in TIER1 with complete FFPE/clinical data match.
  2. - Number of recruited CRC cases in TIER2.

SECONDARY OUTCOMES:
Number of patients triaged in proof-of-concept (POC) clinical trials | 6 months
  Number of CRC cases recruited in TIER3.

OTHER OUTCOMES:
Number of new prognostic and predictive biomarkers | 6 months
  1. - Number of identified/validated new prognostic markers
  2. - Number of identified/validated new predictive markers.
Correlation of new prognostic and predictive biomarkers with clinical outcomes | 6 months
  1. - Correlation between identified biomarkers with therapies response rates (RR).
  2. - Correlation between identified biomarkers with progression-free survival (PFS).
  3. - Correlation between identified biomarkers with overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Marsoni, MD, Principal Investigator — IFOM ETS - The AIRC Institute of Molecular Oncology
Locations (19):
- Italy (14):
  - ASL di Biella - Ospedale degli Infermi, Biella, Biella
  - IRCCS Istituto Clinico Humanitas, Milan, MI
  - Fondazione IRCCS, Istituto Nazionale dei Tumori, Milan, MI
  - Istituto Europeo di Oncologia (IEO), Milan, Mi
  - Niguarda Cancer Center - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Istituto Oncologico Veneto (IOV), Padua, PD
  - Ospedale Santa Maria della Misericordia, Perugia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Pisa
  - AUSL della Romagna - Ospedale Santa Maria delle Croci, Ravenna, Ravenna
  - Istituto di Candiolo - IRCCS, Candiolo, Torino
  - Azienda Ospedaliero Universitaria San Luigi Gonzaga, Orbassano, Torino
  - Ospedale Policlinico San Martino, Genova
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli, Napoli
  - Azienda Ospedaliera Ordine Mauriziano, Torino
- Spain (5):
  - Hospital de Sant Joan Despí Moises Broggi, Barcelona, Barcelona
  - Hospital del Mar - Parc de Salut Mar, Barcelona, Spain
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Spain
  - INCLIVA - Instituto de Investigatión Sanitaria, Valencia, Spain
  - Hospital Moises Broggi, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided